CLINICAL TRIAL: NCT04150081
Title: Endoscopic Versus Surgical Treatment for T1 Colorectal Cancer: a Population-based Cohort Study
Brief Title: Endoscopic Versus Surgical Treatment for T1 Colorectal Cancer
Acronym: EpiT1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, María Pellisé, Principal Investigator. Attending physician Gastroenterology department., Hospital Clinic of Barcelona
Other Study IDs: HCB/2019/0224
Record Dates: First submitted 2019-10-17; First posted 2019-11-04 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer
Keywords: T1 Colorectal Cancer; Early Colorectal Cancer; Endoscopic polypectomy; Oncological Surgery; Lymph node metastasis; Molecular signatures; Disease free survival
MeSH Terms: conditions — Colorectal Neoplasms; Lymphatic Metastasis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Tissue samples. A 10μm slice of the FFPE block will be obtained after manual microdissection of the area with cancer. The molecular study will be carried out in patients who have signed a biobank informed consent prior to the start of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery or Endoscopic treatment — All the patients in the cohort will receive surgery o local (endoscopic) treatment, in some cases additional surgical treatment will be performed after an endoscopic primary treatment. This decision will have been taken based on daily clinical practice and does not represent a study intervention.

SUMMARY:
The implementation of population screening programs for colorectal cancer (CRC) has led to a considerable increase in the prevalence T1 CRC originating on polyps amenable by endoscopy. The benefits of secondary oncological surgery in terms of disease free survival are not well established.

Hypothesis: The characteristics of the individuals and the polyp (endoscopic, histological) should allow us to discriminate T1 CRCs that may benefit from secondary surgery from those that only require local treatment. With the current criteria, the management of patients with T1 CRC is suboptimal since a high proportion of patients are refered for unnecessary surgeries without a clear benefit in terms of survival. Molecular signatures can help to discriminate those patients with good prognosis that do not require secondary surgery nor cancer related follow up.

DETAILED DESCRIPTION:
The primary objective of the study is to compare the effect of oncological surgery versus local treatment for the management of polyps with T1 CRC in relation to disease-free survival and morbi-mortality of the therapeutic procedure. We will also validate molecular signatures in endoscopic samples for the prediction of lymph node metastasis and survival. Methodology: Clinical Study: Retrospective population-based cohort study that will include baseline clinical and follow up data of more than 1400 T1 CRCs in at least 10 Spanish autonomous communities from 2007 to 2017. A centralized pathological review will be carried out by a group of expert pathologists. Inter and intraobserver variability for histological staging will be assessed. A predictive model will be created to discriminate individuals with high probability of receiving surgical and local treatment. For those patients who have a similar probability range, the results in progression-free survival and adverse events will be compared. Translational phase: A 5miRNAs and 8mRNA signature predictive of lymph node metastasis will be assessed in 200 endoscopic samples and related with prognosis.

ELIGIBILITY:
Inclusion Criteria:

- All patients diagnosed with pT1 CRC will be included, regardless of endoscopic features, treatment received and lymph node staging

Exclusion Criteria:

* CRC with other histology than adenocarcinoma
* Patients with hereditary syndromes of CRC (Lynch syndrome, classical familial adenomatous polyposis) or inflammatory bowel disease.
* Synchronous CRC
* Metachronous CRC in the previous 5 years
* Patients with metastatic neoplastic disease at the time of diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Spanish multicenter observational retrospective cohort study where all cases of pT1 CRC will be included from January 2007 to December 2017. Patients will be included both inside and outside the CCR national screening program.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  Evaluate the effect of surgery and local (endoscopic) treatment on overall survival (expressed in months)
Disease free survival | 1 year
  Evaluate the effect of surgery and local (endoscopic) treatment on disease free survival (expressed in months)
Develop a predictive model of the probability of receiving surgical treatment | 1 year
  Determine factors associated with the choice of primary treatment and final treatment (endoscopic, primary surgery or secondary surgery) and to develop a predictive model that allow discriminate individuals with high probability of receiving surgical treatment
Validation of molecular signatures | 2 years
  Evaluate the validity of molecular signatures based on mRNA and miRNA (determined in endoscopic samples) for prediction lymph node metastasis

SECONDARY OUTCOMES:
Prognosis | 1 year
  Determine the prognosis of patients with pT1CRC in relation to the treatment received (local, primary surgery or secondary surgery)
Risk of lymph node metastasis | 1 year
  Evaluate the factors of the individual and the polyp that are associated with lymph node metastasis
Concordance of histological evaluation | 2 years
  Evaluate the inter-intraexplorer concordance of the pathologists for the histological staging criteria.
T1 CRC in screening program | 1 year
  Compare the characteristics of the T1 CRCs diagnosed within a population screening program and outside it.
Proportion of adverse events | 1 year
  Evaluate the proportion of adverse effects after endoscopic or surgical treatment
Sensitivity and specificity of follow-up tests | 1 year
  To evaluate the performances of the different tests (CT, US, blood markers, colonoscopy) during follow up for detecting recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- María Pellisé. MD. PhD., Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Logan RF, Patnick J, Nickerson C, Coleman L, Rutter MD, von Wagner C; English Bowel Cancer Screening Evaluation Committee. Outcomes of the Bowel Cancer Screening Programme (BCSP) in England after the first 1 million tests. Gut. 2012 Oct;61(10):1439-46. doi: 10.1136/gutjnl-2011-300843. Epub 2011 Dec 7. PMID 22156981
- [Background] Williams JG, Pullan RD, Hill J, Horgan PG, Salmo E, Buchanan GN, Rasheed S, McGee SG, Haboubi N; Association of Coloproctology of Great Britain and Ireland. Management of the malignant colorectal polyp: ACPGBI position statement. Colorectal Dis. 2013 Aug;15 Suppl 2:1-38. doi: 10.1111/codi.12262. No abstract available. PMID 23848492
- [Background] Ueno H, Mochizuki H, Hashiguchi Y, Shimazaki H, Aida S, Hase K, Matsukuma S, Kanai T, Kurihara H, Ozawa K, Yoshimura K, Bekku S. Risk factors for an adverse outcome in early invasive colorectal carcinoma. Gastroenterology. 2004 Aug;127(2):385-94. doi: 10.1053/j.gastro.2004.04.022. PMID 15300569
- [Background] Hashiguchi Y, Muro K, Saito Y, Ito Y, Ajioka Y, Hamaguchi T, Hasegawa K, Hotta K, Ishida H, Ishiguro M, Ishihara S, Kanemitsu Y, Kinugasa Y, Murofushi K, Nakajima TE, Oka S, Tanaka T, Taniguchi H, Tsuji A, Uehara K, Ueno H, Yamanaka T, Yamazaki K, Yoshida M, Yoshino T, Itabashi M, Sakamaki K, Sano K, Shimada Y, Tanaka S, Uetake H, Yamaguchi S, Yamaguchi N, Kobayashi H, Matsuda K, Kotake K, Sugihara K; Japanese Society for Cancer of the Colon and Rectum. Japanese Society for Cancer of the Colon and Rectum (JSCCR) guidelines 2019 for the treatment of colorectal cancer. Int J Clin Oncol. 2020 Jan;25(1):1-42. doi: 10.1007/s10147-019-01485-z. Epub 2019 Jun 15. PMID 31203527
- [Background] Benson AB, Venook AP, Al-Hawary MM, Cederquist L, Chen YJ, Ciombor KK, Cohen S, Cooper HS, Deming D, Engstrom PF, Garrido-Laguna I, Grem JL, Grothey A, Hochster HS, Hoffe S, Hunt S, Kamel A, Kirilcuk N, Krishnamurthi S, Messersmith WA, Meyerhardt J, Miller ED, Mulcahy MF, Murphy JD, Nurkin S, Saltz L, Sharma S, Shibata D, Skibber JM, Sofocleous CT, Stoffel EM, Stotsky-Himelfarb E, Willett CG, Wuthrick E, Gregory KM, Freedman-Cass DA. NCCN Guidelines Insights: Colon Cancer, Version 2.2018. J Natl Compr Canc Netw. 2018 Apr;16(4):359-369. doi: 10.6004/jnccn.2018.0021. PMID 29632055
- [Background] Glynne-Jones R, Wyrwicz L, Tiret E, Brown G, Rodel C, Cervantes A, Arnold D; ESMO Guidelines Committee. Rectal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv22-iv40. doi: 10.1093/annonc/mdx224. No abstract available. PMID 28881920
- [Background] Belderbos TD, van Erning FN, de Hingh IH, van Oijen MG, Lemmens VE, Siersema PD. Long-term Recurrence-free Survival After Standard Endoscopic Resection Versus Surgical Resection of Submucosal Invasive Colorectal Cancer: A Population-based Study. Clin Gastroenterol Hepatol. 2017 Mar;15(3):403-411.e1. doi: 10.1016/j.cgh.2016.08.041. Epub 2016 Sep 5. PMID 27609703
- [Background] Hassan C, Zullo A, Risio M, Rossini FP, Morini S. Histologic risk factors and clinical outcome in colorectal malignant polyp: a pooled-data analysis. Dis Colon Rectum. 2005 Aug;48(8):1588-96. doi: 10.1007/s10350-005-0063-3. PMID 15937622
- [Background] Beaton C, Twine CP, Williams GL, Radcliffe AG. Systematic review and meta-analysis of histopathological factors influencing the risk of lymph node metastasis in early colorectal cancer. Colorectal Dis. 2013 Jul;15(7):788-97. doi: 10.1111/codi.12129. PMID 23331927
- [Background] Yoda Y, Ikematsu H, Matsuda T, Yamaguchi Y, Hotta K, Kobayashi N, Fujii T, Oono Y, Sakamoto T, Nakajima T, Takao M, Shinohara T, Fujimori T, Kaneko K, Saito Y. A large-scale multicenter study of long-term outcomes after endoscopic resection for submucosal invasive colorectal cancer. Endoscopy. 2013 Sep;45(9):718-24. doi: 10.1055/s-0033-1344234. Epub 2013 Aug 5. PMID 23918621
- [Background] Lopez A, Bouvier AM, Jooste V, Cottet V, Romain G, Faivre J, Manfredi S, Lepage C. Outcomes following polypectomy for malignant colorectal polyps are similar to those following surgery in the general population. Gut. 2019 Jan;68(1):111-117. doi: 10.1136/gutjnl-2016-312093. Epub 2017 Oct 26. PMID 29074726
- [Background] Ozawa T, Kandimalla R, Gao F, Nozawa H, Hata K, Nagata H, Okada S, Izumi D, Baba H, Fleshman J, Wang X, Watanabe T, Goel A. A MicroRNA Signature Associated With Metastasis of T1 Colorectal Cancers to Lymph Nodes. Gastroenterology. 2018 Mar;154(4):844-848.e7. doi: 10.1053/j.gastro.2017.11.275. Epub 2017 Dec 2. PMID 29199088
- [Background] Backes Y, de Vos Tot Nederveen Cappel WH, van Bergeijk J, Ter Borg F, Schwartz MP, Spanier BWM, Geesing JMJ, Kessels K, Kerkhof M, Groen JN, Wolfhagen FHJ, Seerden TCJ, van Lelyveld N, Offerhaus GJA, Siersema PD, Lacle MM, Moons LMG. Risk for Incomplete Resection after Macroscopic Radical Endoscopic Resection of T1 Colorectal Cancer: A Multicenter Cohort Study. Am J Gastroenterol. 2017 May;112(5):785-796. doi: 10.1038/ajg.2017.58. Epub 2017 Mar 21. PMID 28323275
- [Background] Richards CH, Ventham NT, Mansouri D, Wilson M, Ramsay G, Mackay CD, Parnaby CN, Smith D, On J, Speake D, McFarlane G, Neo YN, Aitken E, Forrest C, Knight K, McKay A, Nair H, Mulholland C, Robertson JH, Carey FA, Steele R; Scottish Surgical Research Group. An evidence-based treatment algorithm for colorectal polyp cancers: results from the Scottish Screen-detected Polyp Cancer Study (SSPoCS). Gut. 2018 Feb;67(2):299-306. doi: 10.1136/gutjnl-2016-312201. Epub 2016 Oct 27. PMID 27789658
- [Background] Overwater A, Kessels K, Elias SG, Backes Y, Spanier BWM, Seerden TCJ, Pullens HJM, de Vos Tot Nederveen Cappel WH, van den Blink A, Offerhaus GJA, van Bergeijk J, Kerkhof M, Geesing JMJ, Groen JN, van Lelyveld N, Ter Borg F, Wolfhagen F, Siersema PD, Lacle MM, Moons LMG; Dutch T1 CRC Working Group. Endoscopic resection of high-risk T1 colorectal carcinoma prior to surgical resection has no adverse effect on long-term outcomes. Gut. 2018 Feb;67(2):284-290. doi: 10.1136/gutjnl-2015-310961. Epub 2016 Nov 3. PMID 27811313
- [Background] Oka S, Tanaka S, Saito Y, Iishi H, Kudo SE, Ikematsu H, Igarashi M, Saitoh Y, Inoue Y, Kobayashi K, Hisabe T, Tsuruta O, Sano Y, Yamano H, Shimizu S, Yahagi N, Watanabe T, Nakamura H, Fujii T, Ishikawa H, Sugihara K; Colorectal Endoscopic Resection Standardization Implementation Working Group of the Japanese Society for Cancer of the Colon and Rectum, Tokyo, Japan. Local recurrence after endoscopic resection for large colorectal neoplasia: a multicenter prospective study in Japan. Am J Gastroenterol. 2015 May;110(5):697-707. doi: 10.1038/ajg.2015.96. Epub 2015 Apr 7. PMID 25848926